CLINICAL TRIAL: NCT04661761
Title: Influence of Two Paraffin Wax Chewing Gums of Different Consistency on the Stimulated Saliva Flow Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-00470; ex20Filippi5
Record Dates: First submitted 2020-12-01; First posted 2020-12-10 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Xerostomia
Keywords: paraffin chewing gum; sialometry; salivary flow rate; mouth dryness
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: Determination of salivary flow rate chewing Paraffin pellets (manufactured by Aurosan GmbH) for 7 minutes. At a later timepoint determination of salivary flow rate chewing Saliva-Check Buffer (manufactured by GC Europe) for 7 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stimulated salivary flow rate (Experimental): stimulated salivary flow rate determined in a crossover design: first using Paraffin Pellets from Aurosan GmbH; thereafter using Chewing wax from the Saliva-Check Buffer from GC Europe
  Interventions: Diagnostic Test: Paraffin Pellets from Aurosan GmbH; Diagnostic Test: Chewing wax from the Saliva-Check Buffer from GC Europe

INTERVENTIONS:
Diagnostic Test: Paraffin Pellets from Aurosan GmbH — 1 to 2 minutes pre-chewing time chewing Paraffin Pellets from Aurosan GmbH, after which the amount of saliva is collected over a period of five minutes. The patient may chew the chewing gum once per second; after each minute the produced amount of saliva is spit in a cup, the whole amount measured after 5 minutes.
Diagnostic Test: Chewing wax from the Saliva-Check Buffer from GC Europe — 1 to 2 minutes pre-chewing time chewing wax from the Saliva-Check Buffer from GC Europe, after which the amount of saliva is collected over a period of five minutes. The patient may chew the chewing gum once per second; after each minute the produced amount of saliva is spit in a cup, the whole amount measured after 5 minutes.

SUMMARY:
The study examines two different chewing gums with regard to consistency and its influence on the result of sialometry

DETAILED DESCRIPTION:
The examination (sialometry) is performed on healthy volunteers. The volunteers must chew on a paraffin gum for seven minutes. After each minute, the amount of secreted saliva is spat into a designated cup and evaluated. This test is performed with Aurosan chewing gum and later with GC Europe chewing gum.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* non-smoker
* no medication

Exclusion Criteria:

* physical or mental illnesses
* smokers
* regular medication intake
* pregnant women
* dementia or persons who are unable to judge or persons with guardianship
* minor test persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2022-04-24 (Actual)

PRIMARY OUTCOMES:
Stimulated salivary flow rate (ml) | at baseline (approx 40 minutes)
  Comparing measurements of stimulated salivary flow rate (ml) after chewing two different chewing gums

SECONDARY OUTCOMES:
Change in consistency of chewing gum | at baseline (7 minutes for each chewing gum)
  Change in consistency (compressive strength, measured in Newton) of the chewing gums for stimulated salivary flow rate measurement over a time period of 7 minutes chewing time

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Filippi, Prof, Principal Investigator — University Center for Dentistry Basel UZB
Locations (1):
- University Center for Dentistry Basel UZB, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No